CLINICAL TRIAL: NCT06619873
Title: A Phase 1, Open-Label, Single-Dose, Randomized, Four-Period Crossover Study to Evaluate the Relative Bioavailability and Food Effect of HRS-8080 in Healthy Subjects
Brief Title: A Phase 1, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of HRS-8080 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-102
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Medication regimen A-D-B-C (Experimental)
  Interventions: Drug: HRS-8080
- Medication regimen B-A-C-D (Experimental)
  Interventions: Drug: HRS-8080
- Medication regimen C-B-D-A (Experimental)
  Interventions: Drug: HRS-8080
- Medication regimen D-C-A-B (Experimental)
  Interventions: Drug: HRS-8080

INTERVENTIONS:
Drug: HRS-8080 — Medication regimen A
  Drug:
  600mg, Old process tablets，NPO
  Medication regimen B
  Drug:
  600mg, New process tablets，NPO
  Medication regimen C
  Drug:
  600mg, New process tablets，PC.，low-fat diet
  Medication regimen D
  Drug:
  600mg, New process tablets，PC.，high-fat diet

SUMMARY:
The study is being conducted to evaluate the relative bioavailability of HRS-8080 in the fasted state in healthy adult subjects and to assess the impact of food on HRS-8080 PK for the Phase 3 capsule in healthy adult.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial.
2. Between 18 and 45 years of age, inclusive
3. Female subjects with weight ≥ 45kg, male subjects with weight ≥50kg, body mass index (BMI) range 19 to 26 kg/m2, inclusive at Screening;
4. Subjects of childbearing potential must agree to take contraceptive measures, and use requested contraceptive measures with their partners from signing the ICF to 6 months after the last dose. Female subjects must have a negative serum pregnancy test within 7 days prior to the first dose, be non-lactating, and agree to avoid egg donation during the treatment period until 6 months after the last dose of the investigational drug;

Exclusion Criteria:

1. Having a significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the Investigator);
2. Having a history of epilepsy, including childhood febrile seizures, loss of consciousness, transient ischemic attack or any condition that may cause seizures, such as cerebrovascular disease, brain injury, stroke or brain cancer, etc.;
3. History of severe infection within the past 30 days, including but not limited to bacteremia, severe sepsis, pneumonia requiring hospitalization
4. History of stomach or intestinal surgery (including cholecystectomy) or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed;
5. Clinically significant findings from medical history, 12-lead ECG, or vital signs;
6. GFR < 90 ml/min/1.73 m2;
7. Having a QTc interval >470 msec for female and >450 msec for male;
8. Positive hepatitis panel (hepatitis B surface antigen and hepatitis C virus antibody) or human immunodeficiency virus (HIV) antibody screens;
9. Having a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator; History of allergy to HRS-8080 or any of its excipients;
10. The use or intent to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including prescription medication, over the counter medication and traditional Chinese medication, within 30 days prior to sreening;
11. The participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to screening;
12. Participated in blood donation within 3 months before screening and donated ≥ 400 mL of blood or ≥ 400 mL of blood loss; Participated in blood donation within 1 month before screening and donated blood volume ≥ 200 mL or blood loss ≥ 200 mL; Those who have received blood transfusions or used blood products within 3 months before screening;
13. Positive test for selected drugs of abuse at Screening;
14. The use of drugs of abuse (including opioids) within3 months of Screening;
15. having a history of alcoholism or heavy smoker within 3 month prior screening; unable to abstain from smoking or alcohol during the trial period;
16. Poor peripheral venous access;
17. The need to follow a special diet and unable to consume the high-fat meal;
18. Pregnant or Breastfeeding;
19. In the opinion of the Investigator or Sponsor, are unsuitable for inclusion in the study;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0 hour-48 hour
AUC0-t | 0 hour-48 hour
AUC0-inf | 0 hour-48 hour

SECONDARY OUTCOMES:
Tmax | 0 hour-48 hour
T1/2 | 0 hour-48 hour
CL/F | 0 hour-48 hour
Vz/F | 0 hour-48 hour

CONTACTS AND LOCATIONS:
Locations (1):
- The Frist Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided